CLINICAL TRIAL: NCT04281914
Title: Reliability and Validity of The Turkish Version of the Functional Assessment of Chronic Illness Therapy - Treatment Satisfaction - General Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Yasin Ekinci, MSc, Hacettepe University
Other Study IDs: GO 19/881
Record Dates: First submitted 2020-02-21; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Satisfaction, Patient
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In the evaluation of the services provided in hospitals in recent years, importance has been given to the measurements based on the perception of the patients. Today, the most frequently used criteria for this purpose are quality of life and patient satisfaction. The general opinion of the experts is that the information obtained with these criteria is valid and reliable.The researchers pointed out that patients who are dissatisfied with the health service provided comply with the recommendations of the healthcare personnel less and thus the primary and secondary preventive services are adversely affected.Although treatment satisfaction is a very important factor in terms of patient adherence to treatment, there is no valid and reliable scale in Turkish to evaluate this factor. This study was carried out to investigate the validity and reliability of The Turkish version of the Functional Assessment of Chronic Illness Therapy - Treatment Satisfaction - General Questionnaire in the patients receiving health care.

ELIGIBILITY:
Inclusion Criteria:

Getting at least 3 sessions of physiotherapy and rehabilitation services, To be at the cooperative level to understand and answer the surveys. Volunteering to participate in the study.

Exclusion Criteria:

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients undergoing physiotherapy and rehabilitation
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 | 30 July 2020